CLINICAL TRIAL: NCT03758339
Title: A Phase 1, Open-label Study of the Absorption, Metabolism, and Excretion of [¹⁴C]-Tucatinib Following a Single Oral Dose in Healthy Male and Female Subjects
Brief Title: A Study of the Absorption, Metabolism, and Excretion of Tucatinib in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cascadian Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONT-380-008
Record Dates: First submitted 2018-11-13; First posted 2018-11-29 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Healthy
MeSH Terms: interventions — tucatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tucatinib (Experimental)
  Interventions: Drug: tucatinib

INTERVENTIONS:
Drug: tucatinib — Single dose of 300 mg of [¹⁴C]-tucatinib containing approximately 150 μCi of [¹⁴C] radioactivity

SUMMARY:
This study will look at how a drug (tucatinib) leaves the body and what happens to tucatinib while it is still in the body. Healthy participants will get one dose of tucatinib by mouth. Patients will be monitored for 8-14 days after they take the dose of tucatinib.

DETAILED DESCRIPTION:
This study will examine the absorption, metabolism, and excretion of tucatinib in healthy individuals. Participants will receive one oral dose of tucatinib and will be followed for 8-14 days after the dose is received.

ELIGIBILITY:
Inclusion Criteria:

* In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital signs measurements, or lab evaluations
* Body mass index (BMI) between 18 and 32 kg/m²
* Weight between 50 and 100 kg
* Females must be of non-childbearing potential
* Males must agree to use contraception

Exclusion Criteria:

* History of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder
* Any condition affecting drug absorption
* History of hypersensitivity or allergy to any drug compound, food, or other substance
* History of alcoholism or drug/chemical abuse within 2 years
* Use of prescription products within 28 days prior to check in
* Use of tobacco- or nicotine-containing products within 3 months prior to check in

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-12-30 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve (AUC) from time 0 to infinity (AUC[0-inf]) | Up to 14 days
  PK outcome parameter for tucatinib, ONT-993, and total radioactivity derived from the whole blood and plasma concentration-time profiles
AUC from time 0 to last quantifiable concentration | Up to 14 days
  PK outcome parameter for tucatinib, ONT-993, and total radioactivity derived from the whole blood and plasma concentration-time profiles
Maximum observed concentration | Up to 14 days
  PK outcome parameter for tucatinib, ONT-993, and total radioactivity derived from the whole blood and plasma concentration-time profiles
Time of maximum observed concentration | Up to 14 days
  PK outcome parameter for tucatinib, ONT-993, and total radioactivity derived from the whole blood and plasma concentration-time profiles
Apparent terminal elimination half-life | Up to 14 days
  PK outcome parameter for tucatinib, ONT-993, and total radioactivity derived from the whole blood and plasma concentration-time profiles
Apparent total clearance | Up to 14 days
  PK outcome parameter for tucatinib derived from the whole blood and plasma concentration-time profiles
Apparent volume of distribution | Up to 14 days
  PK outcome parameter for tucatinib derived from the whole blood and plasma concentration-time profiles
AUC[0-inf] plasma tucatinib/total radioactivity ratio | Up to 14 days
  AUC[0-inf] of plasma tucatinib relative to AUC[0-inf] of plasma total radioactivity
AUC[0-inf] blood/plasma ratio | Up to 14 days
  AUC[0-inf] of whole blood total radioactivity to AUC[0-inf] of plasma total radioactivity
Amount excreted in urine (Aeu) | Up to 14 days
  PK outcome endpoint of tucatinib, ONT-993, and total radioactivity derived from urine collections
Cumulative Aeu | Up to 14 days
  PK outcome endpoint of tucatinib, ONT-993, and total radioactivity derived from urine collections
Percentage excreted in urine (Feu) | Up to 14 days
  PK outcome endpoint of tucatinib and total radioactivity derived from urine collections
Cumulative Feu | Up 14 days
  PK outcome endpoint of tucatinib and total radioactivity derived from urine collections
Renal clearance | Up to 14 days
  PK outcome endpoint of tucatinib derived from urine collections
Amount excreted in feces [Aef] | Up to 14 days
  PK outcome endpoint of total radioactivity derived from feces collection
Cumulative Aef | Up to 14 days
  PK outcome endpoint of total radioactivity derived from feces collection
Percentage excreted in feces [Fef] | Up to 14 days
  PK outcome endpoint of total radioactivity derived from feces collection
Cumulative Fef | Up to 14 days
  PK outcome endpoint of total radioactivity derived from feces collection

SECONDARY OUTCOMES:
Relative abundance of tucatinib and its metabolites eliminated in urine and feces | Up to 14 days
Relative abundance of tucatinib and its metabolites in plasma | Up to 14 days
Incidence of adverse events (AEs) | Up to 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Alex Vo, PhD, Study Director — Cascadian Therapeutics Inc.
Locations (1):
- Covance Clinical Research Unit, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No